CLINICAL TRIAL: NCT03366272
Title: Improvement of Outcome in Elderly Patients or Patients Not Eligible for High-dose Chemotherapy With Aggressive NHL in First Relapse/Progression by Adding Nivolumab to Gemcitabine, Oxaliplatin Plus Rituximab in Case of B-cell Lymphoma
Brief Title: Nivolumab With Gemcitabine, Oxaliplatin + Rituximab in r/r Elderly Lymphoma Patients
Acronym: NIVEAU
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Collaborators: Bristol-Myers Squibb (Industry); Lymphoma Study Association (Other); University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSHNHL 2015-1
Record Dates: First submitted 2017-09-16; First posted 2017-12-08 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Nivolumab; Rituximab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (R)-GemOx (Active Comparator): eight cycles of (R)-GemOx (Gemcitabine 1000 mg/m2, d1, Oxaliplatin 100 mg/m2, d1, Rituximab 375 mg/m2 in case of B-cell lymphoma disease, repeated every 2 wks)
  Interventions: Drug: Rituximab; Drug: Gemcitabine; Device: Oxaliplatin
- Nivo-(R)-GemOx (Experimental): eight cycles of nivolumab (240 mg flatdose) plus (R)-GemOx in 2-wk intervals followed by additional 9 infusions of Nivolumab (480 mg flatdose) in 4-wk intervals as consolidation or up to progression or unacceptable toxicity, whatever occurs first
  Interventions: Drug: Nivolumab; Drug: Rituximab; Drug: Gemcitabine; Device: Oxaliplatin

INTERVENTIONS:
Drug: Nivolumab — eight cycles of nivolumab (240 mg flatdose) plus (R)-GemOx in 2-wk intervals followed by additional 9 infusions of Nivolumab (480 mg flatdose) in 4-wk intervals as consolidation or up to progression or unacceptable toxicity, whatever occurs first
  Arms: Nivo-(R)-GemOx
Drug: Rituximab — eight cycles of R-GemOx in 2-wk intervals
Drug: Gemcitabine — eight cycles of (R)-GemOx in 2-wk intervals
Device: Oxaliplatin — eight cycles of (R)-GemOx in 2-wk intervals

SUMMARY:
This study evaluates the addition of nivolumab to gemcitabine, oxaliplatin plus rituximab in case of B-cell lymphoma

DETAILED DESCRIPTION:
International, multicentre, randomised, open-label, treatment optimisation study, preceded by safety run-in phases conducted for B-cell and T-cell lymphoma separately.

ELIGIBILITY:
Inclusion Criteria:

* patients with first relapse or progression of an aggressive Non-Hodgkin's lymphoma
* all patient >65 years of age or > 18 years if not eligible for neither autologous nor allogeneic stem cell transplantation
* all patient >65 years of age or older than 18 years if HCT-CI score > 2 or patients who underwent prior autologous stem cell transplantation and are not eligible for allogeneic stem cell Transplantation
* All risk groups (IPI 0 to 5)
* Diagnosis of aggressive Non-Hodgkin's lymphoma, based on an excisional biopsy of a lymph node or on an appropriate sample of a lymph node or of an extranodal involvement at initial diagnosis or relapse or Progression. The entities treated in the study will be based on the WHO 2017 classification.
* ECOG 0 - 2
* only one prior chemotherapy regimen including an anthracycline. The last cytotoxic drug must be given at least four weeks before entering the study. Rituximab must be part of the first-line regimen in case of B-cell lymphoma (except for primary CD20- negative lymphoma). Patients may have received prior radiation therapy as part of their first-line therapy
* Men who are sexually active with women of childbearing potential (WOCBP) must not father a child during and up to 6 months after GemOx and up to 12 months after Rituximab and/or Nivolumab. They are advised to do cryoconservation of sperm prior to treatment.
* Written informed consent of the patient
* Patient must be covered by social security system

Exclusion Criteria:

* Already initiated lymphoma therapy after first relapse or progression
* Serious accompanying disorder or impaired organ function
* WBC < 2.5 G/l, Neutrophils < 2 G/l, Platelets < 100 G/l
* Prolongation of QTc interval > 450 ms, demonstrated in one electrocardiogram (done as triplicate). This does not apply for patients with a block of the right and/or left bundle branch.
* Family history for Long QT-Syndrome
* active, known or suspected autoimmune disease
* no requirement for immunosuppressive doses of systemic corticosteroids
* Chronic active hepatitis B or C
* HIV-infection
* Patients with a severe immunodeficiency
* Previous therapy with Nivolumab,Gemcitabine or Oxaliplatin
* Patients with a "currently active" second malignancy other than non-melanoma skin cancer
* CNS involvement of lymphoma
* Persistent neuropathy grade >2
* Pregnancy or breast-feeding women
* Women of childbearing potential
* Active serious infections not controlled by oral and/or intravenous antibiotics or anti-fungal medication
* Any medical condition which in the opinion of the investigator places the subject at an unacceptably high risk for toxicities
* Lymphomas other than those listed in the inclusion criteria notably indolent lymphoma, Mantle cell lymphoma, Burkitt lymphoma, adult T-cell leukemia/lymphoma.
* Persons not able to understand the impact, nature, risks and consequences of the trial (including language barrier)
* Persons not agreeing to the transmission of their pseudonymous data
* Persons depending on sponsor or investigator
* Persons from highly protected Groups
* Allergies and Adverse Drug Reaction History to study drug components
* Participation in another clinical trial with drug intervention within 4 weeks prior to start of the first cycle and during the study. However, participation in a clinical trial of firstline therapy of lymphoma is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
PFS | 1 year
  Progression free survival

SECONDARY OUTCOMES:
CR rate | 4-6 weeks after cycle 8 (each cycle is 14 days)
  complete response rate
PR rate | 4-6 weeks after cycle 8 (each cycle is 14 days)
  partial response rate
ORR rate | 4-6 weeks after cycle 8 (each cycle is 14 days)
  overall response rate
Duration of response | up to 2 years after inclusion of last patient
  Duration of response
Primary Progression rate | up to 2 years after inclusion of last patient
  Rate of Primary progression
Treatment related deaths rate | up to 2 years after inclusion of last patient
  Rate of Treatment related deaths
Relapse rate | up to 2 years after inclusion of last patient
  Rate of relapses
EFS | up to 2 years after inclusion of last patient
  Event free survival
OS | up to 2 years after inclusion of last patient
  Overall survival
Toxicities: rates and grades of adverse events | up to 2 years after inclusion of last patient
  Toxicity: Rates and grades of toxicities will be determined according to CTC-v4.03
Protocol adherence according to number of given chemotherapy cycles | up to 2 years after inclusion of last patient
  Protocol adherence will be determined according to number of chemotherapy cycles
Protocol adherence according to duration of given chemotherapy cycles | up to 2 years after inclusion of last patient
  Protocol adherence will be determined according to duration of chemotherapy cycles
Protocol adherence according to cumulative dose of immunochemotherapy given | up to 2 years after inclusion of last patient
  Protocol adherence will be determined according to cumulative dose of immunochemotherapy given
Protocol adherence according to relative dose of immunochemotherapy given | up to 2 years after inclusion of last patient
  Protocol adherence will be determined according to relative dose of immunochemotherapy given
QoL | up to 1 year after inclusion of last patient
  Quality of Life (QoL) will be assessed by the EQ-5D-5L questionnaire
Biological Parameters according to PD-L1 expression alterations | up to 2 years after inclusion of last patient
  Outcome assessment of response according to PD-L1 expression alterations
Biological Parameters according to PD-1 expression | up to 2 years after inclusion of last patient
  Outcome assessment of response according to PD-1 expression
Biological Parameters according to cell of origin | up to 2 years after inclusion of last patient
  Outcome assessment of response according to cell of origin
Biological Parameters according to 9p24.1 alterations | up to 2 years after inclusion of last patient
  Outcome assessment of response according to 9p24.1 alterations

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Held, Prof, Principal Investigator — Universität des Saarlandes
Locations (77):
- Austria (8):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Innsbruck University Hospital, Innsbruck
  - Kepler Universitätsklinikum GmbH- Med. Campus III, Linz
  - Ordensklinikum Linz - Elisabethinen, Linz
  - Ordensklinikum Linz - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Paracelsus Medical University Salzburg, Salzburg
  - Universitätsklinik für Innere Medizin I, AKH Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (5):
  - INSTITUT JULES BORDET -Hematology, Brussels
  - UNIVERSITE CATHOLIQUE DE LOUVAIN SAINT-LUC - Hematology, Brussels
  - UNIVERSITAIR ZIEKENHUIS GENT - Hematology, Ghent
  - CHU DE LIEGE - Hematology, Liège
  - UNIVERSITE CATHOLIQUE DE LOUVAIN MONT GODINNE - Hematology, Yvoir
- France (18):
  - CHU Côte de Nacre - Service Hématologie Clinique, Caen
  - Hôpital Henri Mondor - Unité "Hémopathies Lymphoïdes" - HDJ 11è, Créteil
  - CHU Dijon - Hôpital d'Enfants - Hématologie Clinique, Dijon
  - CHU de Grenoble - Hôpital Albert Michallon - Hématologie Clinique, Grenoble
  - CH Départemental Vendée - Onco-Hématologie, La Roche-sur-Yon
  - CHRU de Lille - Hôpital Claude Hurriez, Lille
  - CHU de Montpellier - Hématologie Clinique, Montpellier
  - CHU de Nantes - Hôtel Dieu - Hématologie, Nantes
  - Hôpital Necker - Hématologie Clinique, Paris
  - Hôpital Saint Louis - Onco-Hématologie, Paris
  - CHU de Bordeaux - Hôpital Haut Lévêque - Centre François Magendie, Pessac
  - CHU Lyon Sud - Hématologie, Pierre-Bénite
  - Hôpital Pontchaillou - Hématologie, Rennes
  - Centre Henri Becquerel - Hématologie, Rouen
  - Institut de Cancèrologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - IUCT Oncopole - Hématologie, Toulouse
  - CHU Nancy - Hôpital de Brabois - Service d'Hématologie et Médecine Interne, Vandœuvre-lès-Nancy
- Germany (27):
  - Sozialstiftung Bamberg, Bamberg
  - Charité - Universitätsklinikum Berlin, Med. Klinik m. S. Hämatologie, Berlin
  - Vivantes Klinikum am Urban, Klinik für Innere, Hämatologie und Onkologie, Berlin
  - Klinikum Chemnitz, Innere Medizin III, Chemnitz
  - BAG Freiberg-Richter, Jacobasch, Wolf, Illmer, Dresden
  - Gemeinschaftspraxis Dres. Mohm, Prange-Krex, Dresden
  - St. Antonius-Hospital Eschweiler, Klinik für Hämatologie, Eschweiler
  - Universitätsklinikum Essen, Klinik für Hämatologie, Essen
  - Universitätsmedizin Göttingen, Klinik für Hämatologie, Göttingen
  - Universitätsklinikum Haale (Saale), Klinik für Innere Medizin IV, Haale
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum des Saarlandes, Innere Med. I, Homburg
  - Westpfalz-Klinikum, Klinik für Innere Medizin I, Kaiserslautern
  - St. Vincentius Kliniken Karlsruhe, Med. Klinik Abt. 2, Karlsruhe
  - Uni Gießen und Marburg, Klinik für Hämatologie, Marburg
  - Stauferklinikum Schwäbisch Gmünd, Zentrum für Innere Medizin, Mutlangen
  - Klinikum der Universität München, Med. Klinik und Poliklinik III, München
  - Universitätsklinikum Münster, Münster
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Universitätsklinikum Regensburg, Klinik für Innere Medizin III, Regensburg
  - Universitätsmedizin Rostock, Klinik für Hämatologie, Rostock
  - Klinikum Stuttgart, Klinik für Hämatologie, Stuttgart
  - Klinikum Mutterhaus der Borromäerinnen, Med. Abteilung I, Trier
  - Krankenhaus der Barmherzigen Brüder, I. Med. Abteilung, Trier
  - Universitätsklinikum Tübingen, Innere Medizin II, Tübingen
  - Uniklinikum Ulm, Klinik für Innere Medizin III, Ulm
  - Schwarzwald-Baar Klinikum, Innere Medizin II, Villingen-Schwenningen
- The Chaim Sheba Medical Center - Division of Hematology and Bone-Marrow Transplantation, Ramat Gan, Israel
- Netherlands (8):
  - MC Alkmaar, Alkmaar
  - AMC Academisch Medisch Centrum, Amsterdam
  - VUMC, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Maxima Medisch Centrum, Eindhoven
  - MC Leeuwarden Zuid, Leeuwarden
  - Antonius Ziekenhuis, Nieuwegein
  - Radboudumc Nijmegen, Nijmegen
- Poland (9):
  - Szpital Specjalistyczny w Brozowie, Brzozów
  - Oncologic Center, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Swietorkrzyskie Centrum Oncologii, Kielce
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr. 1, Lublin
  - Oncologic Center, Tomaszów Mazowiecki
  - Marie Sklodowska-Curie Institute and Oncology, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- Instituto Português Oncologia - Hematology, Lisbon, Portugal